CLINICAL TRIAL: NCT06367673
Title: Clinical Study to Evaluate the Safety and Efficacy of iPSC -NK Cells Targeting CLL1 or CD33 in Patients With Relapsed/Refractory AML
Brief Title: Natural Killer(NK) Cell Therapy Targeting CLL1 or CD33 in Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Hangzhou Qihanjiyin Biotech Co.,Ltd. (Unknown)
Responsible Party: Principal Investigator, He Huang, Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QH-ZYDC-01
Record Dates: First submitted 2024-04-11; First posted 2024-04-16 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: AML, Adult
Keywords: AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-NK cell therapy in Adult subjects with r/r AML (Experimental)
  Interventions: Biological: iPSC-NK cells

INTERVENTIONS:
Biological: iPSC-NK cells — iPSC-NK cells

SUMMARY:
This is a phase 1, first-in-human (FIH), open-label, multicohort study to evaluate the safety, tolerability and preliminary efficacy of CLL1 or CD33 target Chimeric antigen receptor (CAR) -induced pluripotent stem cells derived NK cells in patients with relapsed/refractory AML

DETAILED DESCRIPTION:
Acute myelogenous leukemia (AML) is a potentially cur-able disease; 70% of newly diagnosed patients achievecomplete remission with first-line therapy, but prognosisworsens for relapsed disease in both pediatric and adultpatients.C-type lectin-like molecule-1 and cluster of differentiation antigen 33 has attracted the researchers' attention due to its high expression in AML while being absent in normal hematopoietic stem cell. Accumulating evidence have demonstrated CLL-1 or CD33 is an ideal target for AML.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old.
* Confirmed diagnosis of r/r AML
* CLL1 or CD33 expression is positive in AML blasts.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤1 and life expectancy greater than 12 weeks.
* Adequate organ and marrow function, as defined below:

  1. Blood creatinine (Cr) ≤ 2 x ULN or calculated creatinine clearance (Cockcroft- Gault formula) ≥ 50 mL/min;
  2. Total bilirubin (TBIL) ≤ 2 x the ULN;
  3. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x ULN;
  4. International normalized ratio (INR) and activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN 6.Females of childbearing potential must have a negative serum pregnancy test. 7.Donor specific antibody (DSA) is negative: MFI <= 2000. 8.Provision of signed and dated informed consent form (ICF).

Exclusion Criteria:

* Allergic to drug used in this study.
* Subjects received any antitumor therapy as follows, prior to first NK infusion:

  a. Systemic steroid therapy within 3 days (except physiological replacement therapy):b. Systemic antitumor therapy within 2 weeks or at least 5 half-lives, whichever is less; c. Radiotherapy within 4 weeks; d. Donor lmphocyte infusion within 6 weeks: e. Intrathecal treatment within 1 week; f CAR-T therapy, CAR-NK therapy, or any other genetically modified cell therapy product within 6 months;
* History of allogeneic stem cell transplantation.
* Received the vaccine within 4 weeks pror to the first infusion andor expected to reuire vaccination from the study period to 12 weeks ater the last intusion
* Active central nervous system Leukemia.
* Acute Promyelocytic Leukemia (APL).

  .History of other malicnant tumors, except for those who have achieved omplete remission more than 5 years after radical treatment without any sions of recurence9. History of central nervous system disease or meningeal involvement such as epilepsy, paralysis, aphasia, stroke, etc
* Active autoimmune diseases.
* Serious cardiovascular and cerebrovascular diseases:a. Severe heart rhythm or conduction abnormalities, corrected OT interval (OTc)>480 ms:h, Aute coronay sndrome conestve heat faur. aortic disection-stroke. or other orade 3 or hioher ardiovasular and cerebrovascular events within 6 months orior to firstinfusiorC, New York Heart Association (NYHA) class l or above congestive heart failure or left ventricular eiection fraction (LVEF <50% in olor Doppler echocardiography,d. Hypertension that cannot be controlled by drug.
* Active pulmonary infection: Sp02 90%: Pulmonary embolism, chronic obstructive pulmonary disease, or interstitial lung disease
* Uncontrolled bacterial, fungal, or viral infection.Known HlV infection, active Hepatitis B (HBV) or Hepatitis C (HCV) infection
* Historv of substance abuse.
* Toxicity induced by previous therapy not recovered to s grade 2(NCI-CTCAE 5.0).15. Large suraical treatment within 4 weeks prior to first infusion, not including diagnostic biopsy.16. Pregnant/breastfeeding women.17. nvestigator-assessed presence of any medical or social issue that are likely to interfere with study conduct or may cause increased risk to subiect

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-04-30 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 28 Days from first dose of iPSC NK cell infusion
  Safety and Tolerability

CONTACTS AND LOCATIONS:
Overall Officials: He Huang, MD, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (1):
- the First Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No